CLINICAL TRIAL: NCT00845741
Title: NGAL Evaluation in ED All-Comers
Brief Title: Neutrophil Gelatinase-associated Lipocalin (NGAL) Evaluation in Emergency Department (ED) All-Comers
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Kyle Fortner, CRA, Biosite, Inc.
Other Study IDs: BSTE-0408
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2010-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to evaluate the NGAL point of care device as an aid in the early risk assessment of AKI (acute kidney injury)in an All-Comers ED population.

DETAILED DESCRIPTION:
This is a multi-center prospective pilot clinical study to assess the utility of the Triage neutrophil gelatinase-associated lipocalin (NGAL) Test as an aid in the early risk assessment for development of acute kidney injury (AKI) (sub clinical minimal changes in creatinine levels to complete failure resulting in kidney replacement therapy) in an all-comers population of patients presenting to the Emergency Department (ED) and designated for hospital admission.. The secondary objectives are to assess the utility of the Triage NGAL Test as an aid in the assessment of AKI severity in patients presenting to the ED, to determine if the combination of Triage NGAL measurements and clinical judgment can improve the early risk assessment for the development of AKI and to correlate Triage NGAL levels to patient outcomes.

Approximately 700 adults presenting to the ED and designated for admission to the hospital will be enrolled. The treating physician will note their preliminary ED diagnosis of AKI vs. no AKI (including prerenal azotemia, non-progressive chronic kidney disease (CKD) and preserved renal function) and their level of confidence in that diagnosis as a percentage following the initial exam.

EDTA anti-coagulated blood samples (for Triage NGAL Test) and blood samples for processing to serum (for Cystatin C test) will be collected and measured for NGAL and Cystatin C levels in all subjects at the following time points:

* immediately upon decision to admit to the hospital from the ED [baseline],
* at 6 and 12 hours after baseline draw
* on days 1, 2 and 3 following admission to the hospital, and
* on the day of hospital discharge (if the subject is hospitalized beyond day 3)

The results of these NGAL and Cystatin C assessments will be blinded to the medical team during the study and will not impact the medical management of the subject.

Blood samples for unblinded standard of care assessment of serum creatinine (analyzed at the hospital's laboratory) will also be obtained:

* in the ED [baseline],
* on days 1, 2 and 3 following admission to the hospital, and
* on the day of hospital discharge (if the subject is hospitalized beyond day 3)

Additional study specific blood samples for blinded assessment of serum creatinine (analyzed at the hospital's laboratory) will also be obtained:

• at 6 and 12 hours after baseline draw

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older;
2. Patients presenting to the ED who have been designated for hospital admission
3. Ability to provide blood samples for baseline NGAL, Cystatin C and creatinine levels either prior to or at admission;
4. Ability to provide written informed consent.

Exclusion Criteria:

1. Known history of marked chronic renal insufficiency (e.g., usual serum creatinine ³ 3.0 mg/dL), on dialysis or RRT (either acute or chronic) or in imminent need of dialysis or RRT at enrollment;
2. Patients with urothelial malignancies;
3. Patients not expected to be admitted and therefore unable to fulfil protocol requirements for blood collection out to day 3 post admission time points
4. Prisoners or other institutionalized or vulnerable individuals;
5. Participation in an interventional clinical study within the previous 30 days;
6. Unlikely to be willing or able to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting to the ED and designated for admission to the hospital will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Development of Acute Kidney Injury (AKI) | 0 to 48hrs after ED presentation

SECONDARY OUTCOMES:
Assess the severity of AKI in patients using the NGAL device and clinical judgement. | 0-48hrs after ED presentation

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Sant'Andrea, Rome, Italy